CLINICAL TRIAL: NCT00990808
Title: A Multiple Dose Study to Investigate the Effect of MK0859 on Lipoprotein Metabolism When Added to Ongoing Statin Therapy in Dyslipidemic Patients
Brief Title: The Effect of MK0859 on Lipoprotein Metabolism in Patients With Dyslipidemia (0859-026 AM3)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-026; 0859-026
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panel A (Experimental): Period 1: atorvastatin + placebo to MK0859; Period 2: atorvastatin + MK0859
  Interventions: Drug: anacetrapib; Drug: Comparator: atorvastatin; Drug: Comparator: placebo to MK0859
- Panel B (Experimental): Period 1: placebo to atorvastatin + placebo to MK0859; Period 2: MK0859 + placebo to atorvastatin
  Interventions: Drug: anacetrapib; Drug: Comparator: placebo to MK0859; Drug: Comparator: placebo to atorvastatin

INTERVENTIONS:
Drug: anacetrapib — [Intervention Name: MK0859] MK0859 100 mg tablet once daily for 8 weeks.
Drug: Comparator: atorvastatin — Atorvastatin 20 mg tablet once daily for 4 weeks in Period 1 and 8 weeks in Period 2.
  Arms: Panel A
Drug: Comparator: placebo to MK0859 — Placebo to MK0859 once daily for 4 weeks.
Drug: Comparator: placebo to atorvastatin — Placebo to atorvastatin once daily for 4 weeks in Period 1 and 8 weeks in Period 2.
  Arms: Panel B

SUMMARY:
This study will investigate the effect of MK0859 on lipoprotein metabolism in patients with dyslipidemia already on statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient's weight has been stable for at least 6 weeks
* Patient is in good health based on medical history, physical exam, and laboratory tests
* Patient has dyslipidemia

Exclusion Criteria :

* Patient has a history of stroke, seizures, or major neurological disorders
* Patient has a history of cancer
* Patient is currently taking any lipid-lowering medications or substances except for statins
* Patient consumes excessive amounts of alcohol or caffeine
* Patient has multiple and/or severe allergies to food or drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Difference in Production Rate (PR) and Fractional Catabolic Rate (FCR) of Low Density Lipoprotein (LDL) apoB100 following treatment with MK0859 and atorvastatin versus atorvastatin alone | 12 weeks

SECONDARY OUTCOMES:
Difference in FCR of LDL apoB100 following treatment with MK0859 versus placebo | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Millar JS, Reyes-Soffer G, Jumes P, Dunbar RL, deGoma EM, Baer AL, Karmally W, Donovan DS, Rafeek H, Pollan L, Tohyama J, Johnson-Levonas AO, Wagner JA, Holleran S, Obunike J, Liu Y, Ramakrishnan R, Lassman ME, Gutstein DE, Ginsberg HN, Rader DJ. Anacetrapib lowers LDL by increasing ApoB clearance in mildly hypercholesterolemic subjects. J Clin Invest. 2015 Jun;125(6):2510-22. doi: 10.1172/JCI80025. Epub 2015 May 11. PMID 25961461
- [Derived] Thomas T, Zhou H, Karmally W, Ramakrishnan R, Holleran S, Liu Y, Jumes P, Wagner JA, Hubbard B, Previs SF, Roddy T, Johnson-Levonas AO, Gutstein DE, Marcovina SM, Rader DJ, Ginsberg HN, Millar JS, Reyes-Soffer G. CETP (Cholesteryl Ester Transfer Protein) Inhibition With Anacetrapib Decreases Production of Lipoprotein(a) in Mildly Hypercholesterolemic Subjects. Arterioscler Thromb Vasc Biol. 2017 Sep;37(9):1770-1775. doi: 10.1161/ATVBAHA.117.309549. Epub 2017 Jul 20. PMID 28729361